CLINICAL TRIAL: NCT00002667
Title: EARLY DETECTION OF SECOND PRIMARY LUNG CANCERS BY SPUTUM CYTOLOGY IMMUNOSTAINING
Brief Title: Early Detection of Second Lung Cancer in Patients With Stage I Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: CDR0000064256; E-5593; SWOG-9437; JHOC-9152; NCI-P95-0067
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Immunoenzyme Techniques

INTERVENTIONS:
Other: cytology specimen collection procedure
Other: immunoenzyme technique
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Using new methods to examine sputum samples for the presence of cancer cells may detect lung cancer earlier.

PURPOSE: Screening trial to study the effectiveness of new methods of examining sputum samples to detect second primary lung cancer in patients with resected stage I non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate whether immunostaining of induced sputum specimens improves the sensitivity and specificity of routine morphologic sputum surveillance to detect second primary lung cancer in patients with previously resected nonsmall cell lung cancer. II. Evaluate which patients are at risk of developing a second primary lung cancer by immunostaining specimens from patients with no morphologic atypia on routine Papanicolaou cytology. III. Make available archived sputum samples and bronchial washings for further analysis of new antibodies and techniques. IV. Evaluate whether analysis of elevations of relevant growth factors in bronchial lavage fluid from patients with positive immunostaining or morphologic atypia increases the accuracy of early detection. V. Evaluate whether quantitation of shed antigens in sputum increases the accuracy of early detection. VI. Evaluate whether the extent of airway obstruction, as measured by the forced expiratory volume, can predict an increased risk of developing lung cancer.

OUTLINE: Screening for Second Primary Lung Cancer. Annual sputum induction for Papanicolaou cytology and immunostaining (using monoclonal antibodies 624H12 and 703D4), with optional pulmonary function tests and fiberoptic bronchoscopy with bronchial washings.

PROJECTED ACCRUAL: 1,100 patients will be entered over 3 years. The sample size will be adjusted based on the rate of positive staining in the first 100 patients. Patients followed at uncertified centers are analyzed separately.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage I (T1-2 N0) nonsmall cell lung cancer curatively resected and in regular follow-up for at least 6 weeks Material available for histologic review At least 1 mediastinal node station sampled or at least 2 years since surgery Any of the following histologies eligible: Squamous cell carcinoma Large cell carcinoma Adenocarcinoma (including bronchoalveolar) No small cell anaplastic component No recurrent disease or second primary No synchronous lung cancer of a different histology Concurrent registration on intergroup protocol I91-0001 allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Cardiovascular: No history of severe hypertension, i.e.: Systolic 200 mm Hg or more Diastolic 120 mm Hg or more No MI within 6 weeks Pulmonary: Available for annual sputum induction and clinical evaluation Clinically able to undergo pulmonary function tests (PFTs) and bronchoscopy Refusal of PFTs or bronchoscopy will not effect eligibility PFTs waived if FEV1/FVC < 65% on prior testing No acute respiratory infection Other: No prior uncontrolled malignancy except nonmelanomatous skin cancer Exceptions for malignancy controlled more than 5 years discretionary

PRIOR CONCURRENT THERAPY: Complete surgical resection required as primary therapy At least 6 weeks since resection, any adjuvant chemotherapy or radiotherapy, or thoracoabdominal surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 1995-10-10 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2004-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Ruckdeschel, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute; Paul A. Bunn, MD, Study Chair — University of Colorado, Denver
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania